CLINICAL TRIAL: NCT06680063
Title: Correlation Between Clinical Assessment and Neurophysiological Assessment in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-CIRB 2023/119.0504-1
Record Dates: First submitted 2024-10-01; First posted 2024-11-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Incomplete Spinal Cord Injury; Spastic Tetraplegia; Spastic Paraplegia; Spinal Cord Injury
Keywords: Spinal cord injury; H-reflex; Spasticity
MeSH Terms: conditions — Quadriplegia; Paraplegia; Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a cross-sectional study that aims to explore the correlation between clinical assessment and neurophysiological assessment in SCI. The clinical outcome assessment are modified-Modified Ashworth scale (m-MAS) and lower extremity motor score. The neurophysiological outcome is H-reflex outcome.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) cause disruption of descending control pathway in spinal cord. The disruption of descending control induce impaired motor and sensory function below the level of injury, as well as the electrical signal from supraspinal pathway. During spinal shock phase, spinal motoneuron become hypoexcitability, as resulting in muscle hypotonicity or flaccidity in clinical manifestation. The spinal motoneuron gradually increase during sub-acute to chronic phase as resulting in development of spasticity in SCI. Development of spasticity is realted to increase of spinal motoneuron excitability, which shown in a decrease in H-reflex latency and increase in Hmax/Mmax ratio. A previous study shown a medium correlation between Hmax/Mmax ratio and MAS in SCI and stroke people. Moreover, the MAS shown a strong correlation with Fugle-meyer score in stroke people. However, it remains unclear in correlation between clinical outcome and neurophysiological outcome assessment of spasticity, and the correlation of spasticity and the motor function in SCI.

This study aims to explore the correlation between clinical assessment and neurophysiological assessment of spasticity in SCI.The clinical outcome assessment are modified-Modified Ashworth scale (m-MAS) and lower extremity motor score (LEMS). The lower extremity motor score is obtained from American Spinal Injury Association (ASIA) imapirement scale. The neurophysiological outcome assessment is H-reflex methode. All particiants who will participated into this study will be assessed the m-MAS, LEMS and H-reflex.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with any level of SCI with age between 18-70 years.
* Onset of injury between 1-30 month.
* Presentation of H-reflex.

Exclusion Criteria:

* Having history of other neurological disease e.g. stroke
* Absent of H-reflex.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal cord injury people from Sirindhorn National Medical Rehabilitation Institute (SNMRI)
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
modified-Modified Ashworth scale | 1 day
  The modified-Modified Ashworth scale is a clinical outcome to evaluate level of spasticity in neurological patient. The MAS consists of 6 grading scale, range from 0 to 5; (i) 0: no increase in muscle tone or normal, (ii) 1: slight increase in muscle tone, with a cathch and release or minimal resistance at the end of the range of motion, (iii) 4: slight increase in muscle tone, manifested as a cathch, followed by minimal resistance through the remainder (less than half) of the range of motion, (iv) 3: a marked increase in muscle tone throughout most of the range of motion, but affected parts still easily moved, (v) 4: considered increase in muscle tone, passive movement difficult, (vi) 4: affected parts rigid in flexion or extension.
Lower extremity motor score | 1 day
  The lower extremity motor score (LEMS) is obtained from American Spinal Injury Association (ASIA) imapirment scale. The ASIA imapirment scale consists of motor, sensory and anorectal examination. This assessment is an standard assessment form for SCI. The lower extremity motor score assess 5 key lower extremity muscles. which are hip flexors, knee extensors, ankle plantar flexors, ankle dorsiflexors and long toe extensors. These 5 key muscles represent motor recovery throughout myotome of the body. Grading of this assessment range from 0 to 5, according to mannual muscle testing grading system.
Soleus H-reflex | 1 day
  A most reliable are for assess spinal motoneuron excitability is soleus H-reflex. The stimulation electrode place over the popletial fossa to stimulate tibial nerve. Two disposal surface electrode place over 1/3 of lower leg which is over the soleus muscle. Data from the assessment are H-reflex latency, H-reflex amplitude, M-wave response amplitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Nakhon Pathom, Salaya, Thailand